CLINICAL TRIAL: NCT07246031
Title: An Open-Label, Single-Arm, Phase Ⅱb Clinical Study of BPC2001 for the Prevention of Acute Graft-Versus-Host Disease Following Haploidentical Stem Cell Transplantation
Brief Title: BPC2001 for the Prevention of Acute Graft-Versus-Host Disease Following Haploidentical Stem Cell Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioPhoenix Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BPC2001-01
Record Dates: First submitted 2025-09-22; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Graft -Versus-host-disease; aGVHD; Haploidentical Stem Cell Transplantation; cGVHD
Keywords: aGvHD; Haplo-SCT; BPC2001; BioPhoenix; KRN-7000
MeSH Terms: conditions — Graft vs Host Disease | interventions — KRN 7000

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safety run-in and Expansion (Experimental): Safety Run-in Phase:
  Up to 2 cohorts of at least 3 subjects will be enrolled in the Safety Run-in Phase. The Safety Run in Phase will enroll at least 6 subjects in total. Initially, 3 subjects will be enrolled, treated, and assessed for the dose-limiting toxicity (DLT).
  Expansion Phase:
  Once a dose/schedule with an acceptable safety/PK profile is determined by the SRC, enrollment will continue to the Expansion Phase. The Expansion Phase will enroll 44 subjects. The dose of BPC2001 will be tentatively 100 μg/kg on a weekly basis for 6 doses, and the specific dose and/or schedule will be determined by the SRC based on the data of the Safety Run-in Phase.
  Interventions: Drug: BPC-2001

INTERVENTIONS:
Drug: BPC-2001 — Subjects will receive 6 weekly doses of BPC2001, 100 μg/kg via IV administration after completion of Haplo-SCT.
  Other Names: KRN-7000

SUMMARY:
A Phase IIb open label study evaluates the safety and efficacy of repeat doses of BPC2001 in combination with standard of care treatment for the prevention of acute graft-vs-host-disease (aGvHD) in subjects following Haploidentical Stem Cell Transplantation (Haplo-SCT).

DETAILED DESCRIPTION:
This is an open-label, single center, single-arm study to evaluate six weekly doses of BPC2001 in combination with standard of care treatment (Beijing Protocol) for the prevention of aGvHD in subjects following Haplo-SCT. The study includes a Safety Run-in Phase to assess the safety and tolerability of 30 days DLT after the first dose of BPC2001 followed by an Expansion Phase in which the efficacy of 6 weekly doses of BPC2001 in addition to standard of care for GvHD prophylaxis will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ages ≥18 and ≤ 65 years.
2. Before the start of the trial, the subject or his/her guardian is sufficient to understand and voluntarily sign the written informed consent form (ICF).
3. Subjects have a hematologic malignancy as defined below and are considered candidates for haplo-SCT:

   1. Acute leukemia with morphologic complete remission (acute myelogenous leukemia [AML] or acute lymphoblastic leukemia [ALL]);
   2. Myelodysplastic syndrome (MDS), chronic myelomonocytic leukemia (CMML), or myeloproliferative neoplasm (MPN) with < 10% blasts in the bone marrow.
4. Organ function tolerated for transplantation:

   1. Cardiac function: Left ventricular ejection fraction at rest ≥ 45%;
   2. Liver function: Total bilirubin < 1.5 × upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 × ULN. Subjects who have been diagnosed with Gilbert's syndrome or malignant disease involvement are allowed to have a total bilirubin value > 1.5 × ULN;
   3. Serum creatine < 2 mg/dL or estimated creatinine clearance > 50 mL/min calculated using the Cockcroft-Gault equation；
   4. Pulmonary function tests (PFTs): diffusing capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin) and/or forced expiratory volume in 1 second (FEV1) ≥ 50%.
5. Subject is suitable for myeloablative haplotype related donor transplant.
6. Subject is suitable for receiving first alloHSCT.
7. The transplant donor must meet the following criteria:

   1. Donor ages > 30 years; If the donor ages is equal to or less than 30 years, the donor should be female for male subject;
   2. High-resolution typing of human leukocyte antigen (HLA)-A, -B, -C, DR, and DQ are matched at least 5/10;
   3. Meet the criteria for peripheral blood stem cell (PBSC) donation;
   4. Donor's specific antibodies are negative, <2,000 MFI.
8. Source of allografts: using G-CSF as the mobilizing agent to mobilize PBSC transplant; bone marrow or cord blood is not allowed.
9. Karnofsky Performance Status (KPS) score ≥ 60 points.
10. Is a Candidate for anti-GvHD prophylaxis, including ATG, calcineurin inhibitor (CsA or tacrolimus [FK 506]) in combination with MTX and MMF.
11. Female subjects of childbearing potential must have a negative serum pregnancy test prior to enrollment and must have agreed to use a double barrier method of contraception from the time of signing the ICF to 90 days after the last dose of investigational drug.
12. Male subjects must agree to use effective contraception from the time of signing the ICF to 90 days after the last dose of investigational drug.

Exclusion Criteria:

Any subjects who meet any of the following criteria will be excluded from study entry:

1. Has had any other prior organ transplantation.
2. Planned use of any additional or alternative drugs for GvHD prophylaxis than listed in the inclusion criteria.
3. Has had received an investigational drug within 4 half-lives or within 14 days prior to HSCT, whichever is longer; or plans to participate in another clinical study prior to completion of all scheduled evaluations in this clinical study.
4. Has other malignancies that are not controlled.
5. Has evidence of active central nervous system (CNS) disease.
6. Patients with uncontrolled active bacterial, viral, or fungal infections.
7. Known history of human immunodeficiency virus (HIV) or positive HIV antibody test.
8. Hepatitis B virus surface antigen (HBsAg) or hepatitis B virus core antibody (HBcAb) is positive, and the hepatitis B virus (HBV) DNA in peripheral blood is above the limit of quantification; or hepatitis C virus (HCV) antibody and peripheral HCV RNA are positive; or the syphilis TRUST test is positive.
9. Pregnant or lactating females.
10. Has undergone major surgery within 1 month prior to the first dose of investigational drug.
11. In the opinion of the investigator, the subject has any other medical condition that renders the subject unsuitable for participation in the study.
12. Has a history of uncontrolled autoimmune disease or on active treatment.
13. Vaccinated with live or attenuated vaccine within 4 weeks prior to the first dose of investigational drug.
14. History of myocardial infarction, unstable angina, acute coronary syndrome, congestive heart failure (New York Heart Society classification ≥ class Ⅲ), or clinically significant arrhythmia within 6 months prior to receiving the investigational drug.
15. Plan to use prophylaxis donor lymphocyte infusion (DLI) therapy.
16. The transplant donor is the subject's mother or collateral relative.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2027-11-02 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Grades II-IV aGVHD | Day 100 after the last infusion of stem cell
  To assess the incidence of Grades II-IV aGvHD by Day 100 (D100) after the last infusion of stem cell (the Mount Sinai aGvHD International Consortium [MAGIC] criteria)
AE of BPC2001 in addition to the graft-versus-host disease (GvHD) prophylaxis regimen | 1 year post-transplant
  Incidence, nature, and severity of treatment-emergent adverse events (AEs)
SAE of BPC2001 in addition to the graft-versus-host disease (GvHD) prophylaxis regimen | 1 year post-transplant
  Incidence, nature, and severity of serious adverse events (SAEs)
Lab test values of BPC2001 in addition to the graft-versus-host disease (GvHD) prophylaxis regimen | 1 year post-transplant
  Incidence, nature, and severity of laboratory test values (complete blood count, serum chemistry test, coagulation test and urinalysis)
Vital sign of BPC2001 in addition to the graft-versus-host disease (GvHD) prophylaxis regimen | 1 year post-transplant
  Incidence, nature, and severity of vital sign measures including temperature, blood pressure (systolic/diastolic), pulse, and respiratory rate
Graft failure of BPC2001 in addition to the graft-versus-host disease (GvHD) prophylaxis regimen | 1 year post-transplant
  Incidence, nature, and severity of graft failure

SECONDARY OUTCOMES:
Grades II-IV aGVHD | Day 180 post-transplant
  Acute GVHD will be graded and assessed within 180 days post-transplant
Total and moderate-severe cGvHD | Day 180 and 1 year post-transplant
  Incidence of total and moderate-severe cGvHD assessment
Non-relapse Mortality (NRM) Rates | Day 100, Day 180 and 1 year post-transplant
  The probability of mortality not preceded by relapse of the underlying malignancy will be estimated
Disease-free Survival (DFS) | Day 180 and 1 year post-transplant
  The probability of survival without relapse of the underlying malignancy will be estimated
GvHD-free, Relapse Free Survival (GRFS) | Day 180 and 1 year post-transplant
  The probability of survival without relapse of the underlying malignancy, without severe (grades 3-4) acute GVHD, and without chronic GVHD requiring systemic immunosuppression will be estimated
Overall Survival (OS) | Day 180 and 1 year post-transplant
  The probability of survival will be estimated
PK Profile_Cmax after a single dose of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: maximum observed concentration (Cmax) after a single dose
PK Profile_Tmax after a single dose of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: time to maximum concentration (Tmax) after a single dose
PK Profile_AUC0-t after a single dose of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: area under the concentration versus time curve from time 0 to the time point of the last measurable concentration (AUC0-t) after a single dose
PK Profile_AUC0-inf after a single dose of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: area under the concentration versus time curve from time 0 extrapolated to infinite (AUC0-inf) after a single dose
PK Profile_t1/2 after a single dose of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: terminal half-life (t1/2) after a single dose
PK Profile_CL after a single dose of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: clearance (CL) after a single dose
PK Profile_Vd after a single dose of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: volume of distribution (Vd) after a single dose
PK Profile_Cmax after multiple doses of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: Cmax after multiple doses
PK Profile_Tmax after multiple doses of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: Tmax after multiple doses
PK Profile_AUC0-t after multiple doses of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: AUC0-t after multiple doses
PK Profile_AUC0-inf after multiple doses of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: AUC0-inf after multiple doses
PK Profile_t1/2 after multiple doses of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: t1/2 after multiple doses
PK Profile_Ctrough after multiple doses of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: trough concentration (Ctrough) after multiple doses
PK Profile_CLss after multiple doses of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: clearance at steady state (CLss) after multiple doses
PK Profile_Vss after multiple doses of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: volume of distribution at steady state (Vss) after multiple doses
PK Profile_ARCmax after multiple doses of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: accumulation factors ARCmax after multiple doses
PK Profile_ARAUC after multiple doses of BPC2001 | Day 0 through Day 35
  To calculate the PK parameters of the total drug and free drug (if feasible) in the plasma sample, including but not limited to: ARAUC after multiple doses

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Mo, PhD, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 7.General Office of National Health Commission. Clinical Application Management Standards for Allogeneic Hematopoietic Stem Cell Transplantation Technology (2022 Edition).
- [Background] Ciurea SO, Al Malki MM, Kongtim P, Fuchs EJ, Luznik L, Huang XJ, Ciceri F, Locatelli F, Aversa F, Castagna L, Bacigalupo A, Martelli M, Blaise D, Ben Soussan P, Arnault Y, Handgretinger R, Roy DC, O'Donnell PV, Bashey A, Solomon S, Romee R, Gayoso J, Lazarus HM, Ballen K, Savani BN, Mohty M, Nagler A. The European Society for Blood and Marrow Transplantation (EBMT) consensus recommendations for donor selection in haploidentical hematopoietic cell transplantation. Bone Marrow Transplant. 2020 Jan;55(1):12-24. doi: 10.1038/s41409-019-0499-z. Epub 2019 Mar 4. PMID 30833742
- [Background] Wang Y, Chang YJ, Xu LP, Liu KY, Liu DH, Zhang XH, Chen H, Han W, Chen YH, Wang FR, Wang JZ, Chen Y, Yan CH, Huo MR, Li D, Huang XJ. Who is the best donor for a related HLA haplotype-mismatched transplant? Blood. 2014 Aug 7;124(6):843-50. doi: 10.1182/blood-2014-03-563130. Epub 2014 Jun 10. PMID 24916508
- [Background] Duramad O, Laysang A, Li J, Ishii Y, Namikawa R. Pharmacologic expansion of donor-derived, naturally occurring CD4(+)Foxp3(+) regulatory T cells reduces acute graft-versus-host disease lethality without abrogating the graft-versus-leukemia effect in murine models. Biol Blood Marrow Transplant. 2011 Aug;17(8):1154-68. doi: 10.1016/j.bbmt.2010.11.022. Epub 2010 Dec 8. PMID 21145405
- [Background] Socie G, Blazar BR. Acute graft-versus-host disease: from the bench to the bedside. Blood. 2009 Nov 12;114(20):4327-36. doi: 10.1182/blood-2009-06-204669. Epub 2009 Aug 27. PMID 19713461
- [Background] 2. Hematology Branch Stem Cell Application Group of Chinese Medical Association. Expert Consensus on Diagnosis and Treatment of Acute Graft-versus-Host Disease After Allogeneic Hematopoietic Stem Cell Transplantation (2024 Edition). Chinese Journal of Hematology. 2024;45(6):525-533.
- [Background] 1. Huang Xiaojun. Haploidentical Hematopoietic Stem Cell Transplantation Beijing Protocol, Chinese Journal of Organ Transplantation. 2017;38(2): 65-68.